### **Infant and Child European Cryoablation Project**

ClinicalTrials.gov study ID: 18BB37



**CONFIDENTIAL** 

# 16+/Young Person Assent form

Date of most recent review: 16th November 2020

Version 2 16/11/2020 1

## **Infant and Child European Cryoablation Project**

ClinicalTrials.gov study ID: 18BB37



#### **CONFIDENTIAL**

### **16+/YOUNG PERSON CONSENT FORM**

| | Please In | | | oxes |
|---|---|---|---|---|
| 1. | I confirm that I have read and understand the information sheet(s) dated 05/10/2018 version 1, for the above study, have been informed of the nature, significance, implications and risks associated with it and have had the opportunity to ask questions. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without his/her medical care or legal rights being affected. | | | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible physicians or authorised persons from sponsor organisation, regulatory authorities or hosting organisations where it is relevant to my/my child's taking part in research. I give permission for these individuals to have access to his/her records | | | |
| 4. | I agree to take part in the above study. | | | |
| 5. | i. I agree that I might be contacted in the future for a long-term follow-up | | | |
| Name of Patient | | Date | Signature | |
| No | and of name on taking concept | | | |
| Name of person taking consent (if different from Investigator) | | | | |
| <u>,-</u> | , | | | |
| Na | me of Investigator | | | |
| Na | me of Interpreter (if applicable) | | | |

1 copy for patient, 1 for researcher, 1 copy to be kept with hospital notes

Version 2 16/11/2020 2